CLINICAL TRIAL: NCT05228379
Title: Small Bowel Capsule Endoscopy: Experience From a Single Large Tertiary Care Centre
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AIG/IEC-BH&R 17/08/2021-02
Record Dates: First submitted 2022-01-03; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Small Bowel Disease; Small Bowel Ulcers; Capsule Endoscopy; Small Bowel Tumor
Keywords: capsule endoscopy; small bowel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Small Bowel Capsule Endosocopy — A wireless capsule is ingested by the patient. It moves passively along with the peristaltic movements to capture images of the small intestine. The images are processed and recorded by data recorder worn on a belt. The recorded images are downloaded and analyzed by the computer software.

SUMMARY:
Examination of the small bowel has been considered a challenge for several anatomical (i.e. distance from external orifices, length) and physiological (i.e. active peristalsis) reasons. Conventional techniques of endoscopy are limited by length while radiologic examinations, such as barium studies, are insensitive for evaluating small bowel pathology. An ingestible miniature camera device capable of obtaining images of the whole small intestine was developed due to a need for the exploration of this "final frontier". The purpose of this article is to review and share our institution's results using small bowel capsule endoscopy, with special reference to the existing literature.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Examination of the small bowel (SB) has been considered a challenge for several anatomical (i.e. distance from external orifices, length) and physiological (i.e. active peristalsis) reasons. Conventional techniques of endoscopy are limited by length while radiologic examinations, such as barium studies, are insensitive for the evaluation of pathology in the SB. An ingestible miniature camera device capable of obtaining images of the whole small intestine was developed due to a need for the exploration of this "final frontier". Video capsule endoscopy (CE) is a breakthrough in medical history for noninvasive imaging of the entire small intestine. It was first introduced in 2000, and since then more than 700 studies have been published, which is indicative of its ease and the widespread acceptance of this new diagnostic tool. A wide range of uses for CE has been reported in the literature, but the majority of the studies have aimed to evaluate the cause of obscure gastrointestinal bleeding (OGIB).
2. RATIONALE The purpose of this article is to review and share our institution's experience using small bowel CE, with special reference to the existing literature. Most published reports on capsule endoscopy are limited to small group of patients.
3. STUDY OBJECTIVES 3A. Primary Objective- To study the indications and diagnostic yield of capsule endoscopy.

3B. Secondary Objective- To study the gastric emptying time, small bowel transit time and findings visualized with capsule endoscopy.

4. STUDY POPULATION This observational retrospective study will be conducted in AIG Hospitals, Hyderabad. All patients who underwent capsule endoscopy till 30 June, 2021 will be enrolled in the study.

5. DESIGN AND DURATION OF THE STUDY- It will be a retrospective observational study.

6. METHODOLOGY

6a. SUBJECT RECRUITMENT - All patients who underwent capsule endoscopy in our hospital till 30 June, 2021 will be enrolled in the study.

6b. RANDOMIZATION AND BLINDING- N/A

6c. STUDY METHODS- This observational study will be conducted after obtaining ethical clearance from institutional human ethical committee. All patients who underwent capsule endoscopy till date will be enrolled in the study.

6d. STUDY PROCEDURE- The data will be entered in Microsoft excel sheet and analysed ' 6e. METHODS OF ASSESSMENT- The following variables will be noted. A. Age of the patient B. Indications of the procedure C. Pre-Existing illness D. Gastric Emptying time E. Small Bowel transit time F. Capsule Retention G. Findings visualized on capsule endoscopy study

6e. STOPPING OR DISCONTINUATION CRITERIA- N/A

7. SAMPLE SIZE CALCULATION- The sample size will include all patients who underwent capsule endosocopy till 30th June 2021 in AIG hospitals Hyderabad.

8. STATISTICAL ANALYSIS- Data will be expressed as median and percentile values (5th, 25th, 75th and 95th percentiles). The upper limit of normal will be defined as the 95th percentile of expected values. P≤0.05 will be considered statistically significant.

9. ETHICAL JUSTIFICATION OF THE STUDY Small Bowel Capsule endoscopy is a safe and effective procedure for diagnosis of small bowel disorders. It is especially helpful in finding the cause for obscure gastro-intestinal bleed. There is lack of large studies on diagnostic yield and other visualized findings. This study aims to share our institution's results using small bowel CE, with special reference to the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent capsule endoscopy in AIG Hospitals Hyderbad till 30 June, 2021 will be enrolled in the study.

Exclusion Criteria:

* Patients in whom capsule was unable to reach caecum.

Ages: 6 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes patients who underwent capsule endoscopy from Jan 2013 till 30 June, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1157 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Indications for doing capsule endoscopy procedure | 8-9 years
  The study will help find the various indications for doing capsule endoscopy for small bowel diseases.

SECONDARY OUTCOMES:
Findings visualized on capsule endoscopy. | 8-9 years
  The study will help in knowing the various findings visualized on capsule endoscopy.
Diagnostic yield of capsule endoscopy | 8-9 years
  he study will help find the diagnostic yield of capsule endoscopy for various small bowel diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Singla, MBBS, MD, DM, Principal Investigator — Consultant Gastroenterologist

IPD SHARING:
Plan to Share IPD: Undecided
It's yet undecided.

REFERENCES:
- [Result] Goenka MK, Majumder S, Kumar S, Sethy PK, Goenka U. Single center experience of capsule endoscopy in patients with obscure gastrointestinal bleeding. World J Gastroenterol. 2011 Feb 14;17(6):774-8. doi: 10.3748/wjg.v17.i6.774. PMID 21390148
- [Result] Yung DE, Robertson AR, Davie M, Sidhu R, McAlindon M, Rahman I, Patel P, Sinha L, Mason S, Brzeszczynska J, Douglas S, Plevris JN, Koulaouzidis A. Double-headed small-bowel capsule endoscopy: Real-world experience from a multi-centre British study. Dig Liver Dis. 2021 Apr;53(4):461-466. doi: 10.1016/j.dld.2021.01.017. Epub 2021 Feb 8. PMID 33574013
- [Result] Flemming J, Cameron S. Small bowel capsule endoscopy: Indications, results, and clinical benefit in a University environment. Medicine (Baltimore). 2018 Apr;97(14):e0148. doi: 10.1097/MD.0000000000010148. PMID 29620627
- [Result] Kav T, Bayraktar Y. Five years' experience with capsule endoscopy in a single center. World J Gastroenterol. 2009 Apr 28;15(16):1934-42. doi: 10.3748/wjg.15.1934. PMID 19399924